CLINICAL TRIAL: NCT06096623
Title: The Care Tracker Study: Using Patient-Reported Data to Address Racial Disparities in Cancer Treatment Delay
Brief Title: The Care Tracker Study: Using Patient-Reported Data to Address Racial Disparity in Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC2315
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Breast Cancer; Colorectal Cancer
Keywords: patient-reported outcome; electronic; health equity; electronic survey; treatment delay
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- electronic patient-reported outcome (ePRO) questionnaires. (Experimental): Subjects with colon or breast carcinoma will respond to weekly electronic patient-reported outcome (ePRO) questionnaires.
  Interventions: Behavioral: Weekly Survey

INTERVENTIONS:
Behavioral: Weekly Survey — Subjects will respond to Electronic patient-reported outcome (ePRO) every week for 8 weeks.

SUMMARY:
This study assesses the feasibility and acceptability of a brief electronic patient-reported outcome (ePRO) tool that allows patients to self-identify impending delays. The risk of treatment delays according to tumor type and race will be measured by both ePRO and electronic health record (EHR) tools. Data from this study and the association of social determinants of health could be useful to flag patients at risk of delay and due timely intervention for modifiable treatment barriers. The prediction of the risk of treatment delay will be helpful to design another study using electronic tracking systems to prevent cancer treatment delays. The long-term goal of this research is to alert care teams when patients may be at risk of treatment days and to help patients get treatment faster. It was planned to enroll a total of 240 subjects with newly diagnosed cancer. Sixty colorectal and 180 breast cancer patients will be included.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

1. Male and female patients of age >18 years.
2. Pathologic diagnosis of breasts or colorectal cancer within 6 weeks (42 days) prior to the enrollment date.
3. Have not yet initiated cancer treatment on the date of enrollment.
4. Indicate intent to receive cancer treatment at the University of North Carolina.

Exclusion Criteria:

1. Patient unwilling or unable to receive electronic survey links via email or text link on a mobile device, tablet, laptop, or desktop computer.
2. Patient unwilling or unable to provide verbal or signed consent to participate.
3. Patient cannot read and speak English.
4. Patients who do not have email access or a smartphone are able to receive Short Message/Messaging Service (SMS) text messages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Electronic patient-reported outcome (ePRO) | Baseline to 56 days post-enrollment
  Feasibility of Electronic patient-reported outcome (ePRO) will be assessed as the proportion of subjects who responded to at least 4 out of offered 8 weekly ePRO.
Electronic patient-reported outcome (ePRO) confirming treatment initiation | Baseline to 56 days post-enrollment
  Electronic patient-reported outcome (ePRO) confirming treatment initiation will be measured as the proportion of subjects who responded to at least one of the offered weekly ePRO) surveys.

SECONDARY OUTCOMES:
Delayed Treatment | Baseline to 56 days post-enrollment
  Treatment Delay will be measured as the proportion of subjects not receiving ePRO-reported treatment.
  If a subject reports on any weekly survey that they have started a treatment for their cancer, selected from a defined list of cancer treatment types this will be considered receiving treatment. Diagnostic procedures, imaging tests, and other medical interventions will not be considered receiving treatment. Patients who respond to surveys indicating no treatment throughout the 56 days of study participation, those who report treatment at a timepoint >56 days from pathologic-confirmed diagnosis, as well as those who do not respond to surveys, will be considered as not receiving treatment for this endpoint.
Time to ePRO-reported treatment | Baseline to 56 days post-enrollment
  Time to ePRO-reported treatment will be assessed as the time from the first documented pathologic confirmation of malignancy (or imaging evidence if biopsy was not obtained) to the first day of the week in which the patient reports receiving treatment as per.
  Surveys are completed weekly; thus, the date of treatment is assumed to be the first day of the week in which the patient completes the survey and reports treatment initiation. For instance, if a patient completes a survey on day 32, reporting that they received treatment in the previous week, their date of treatment initiation is assumed to be day 26.
Proportion of treatment delay | Baseline to 56 days post-enrollment
  The proportion of treatment delay will be defined as days between the first documented pathologic confirmation of malignancy to the first therapeutic intervention longer than 56 days divided by the total number of consented patients. Dates will be identified by the study team using a structured abstraction form from either outside medical records captured in the EPIC or UNC EPIC records.
Time to treatment in days | Baseline to 180 days post-enrollment
  Time to treatment in days will be assessed as days between the first documented pathologic confirmation of malignancy to the first therapeutic intervention. Dates will be identified by the study team, using a structured abstraction form from either outside medical records captured in the EPIC or other medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Reeder-Hayes, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials